CLINICAL TRIAL: NCT06080620
Title: Treatment Selection and Efficacy of Locally Advanced Breast cancer-a Prospective Randomized Controlled Study
Brief Title: The Choice of Treatment Methods and Efficacy of LABC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-LABC study
Record Dates: First submitted 2023-09-21; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Locally Advanced Breast Cancer
Keywords: Locally Advanced Breast Cancer; prognosis
MeSH Terms: interventions — Mastectomy, Modified Radical; Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: The plan for Group A (experimental group) is "surgery+systematic treatment"; The plan for Group B (control group) is "neoadjuvant therapy+surgery+systematic treatment".
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Surgery+systematic treatment
  Interventions: Procedure: Modified radical mastectomy for breast cancer; Procedure: Systematic treatment
- Group B (Active Comparator): Neoadjuvant therapy+surgery+systematic treatment
  Interventions: Procedure: Modified radical mastectomy for breast cancer; Procedure: neoadjuvant therapy; Procedure: Systematic treatment

INTERVENTIONS:
Procedure: Modified radical mastectomy for breast cancer — Modified radical mastectomy for breast cancer
Procedure: neoadjuvant therapy — neoadjuvant chemotherapy（Drugs：" Doxorubicin""Paclitaxel""Albumin paclitaxel""Cyclophosphamide"）, endocrine therapy（Drugs："Toremifen""Zoladex""Aromatase inhibitors"）, targeted therapy（Drugs："trastuzumab""Pertuzumab"）
  Arms: Group B
Procedure: Systematic treatment — chemotherapyDrugs：" Doxorubicin""Paclitaxel""Albumin paclitaxel""Cyclophosphamide"）, endocrine therapy（Drugs："Toremifen""Zoladex""Aromatase inhibitors"）, targeted therapy（Drugs："trastuzumab""Pertuzumab"），radiotherapy（"Yikeda Versa HD linear accelerator""Varian Trilogy linear accelerator"）

SUMMARY:
The goal of this clinical trial is to compare the therapeutic effects of chemotherapy followed by surgery and surgery followed by chemotherapy in patients with locally advanced breast cancer（LABC). Patients with LABC will be randomly divided into two groups, each receiving chemotherapy followed by surgery or surgery followed by chemotherapy. The main comparison was between the disease-free survival (DFS) of two groups of patients, with the secondary study endpoint being overall survival (OS); Five year survival; Local recurrence or distant metastasis rate.

DETAILED DESCRIPTION:
Local advanced breast cancer was enrolled in the Department of Breast Surgery of Peking Union Medical College Hospital and Beijing Cooperation Hospital according to the criteria for patient inclusion. It is estimated that 50 patients will be enrolled. Randomly divide patients into two groups. The plan for Group A (experimental group, 25 cases) is "surgery+systematic treatment"; The plan for Group B (control group, 25 cases) is "neoadjuvant therapy+surgery+systematic treatment". Based on the previously obtained patient personal information, treatment related information, tumor tissue/blood sample test results, statistical analysis was conducted to explore the impact of different treatment strategies for locally advanced breast cancer on the survival and prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 year old female
2. Patients with locally advanced breast cancer (stage IIIb - IIIc) first diagnosed;
3. Clinical diagnosis of breast cancer, or puncture pathology suggests breast cancer;
4. After evaluation by experienced clinical physicians, the patient's tumor has the possibility of surgical resection. Specific evaluation indicators include ultrasound assessment of the tumor not surrounding the axillary vein;
5. Accept treatment plans including surgery, radiotherapy, and chemotherapy;
6. Volunteer to participate in clinical research and sign an informed consent form;
7. Willing to undergo follow-up and complete quality of life (EQ-5D series scale and FACT-B scale) and postoperative psychological status (Anxiety/Depression Self Rating Scale) assessments;

Exclusion Criteria:

1. Patients under 18 years old or over 70 years old;
2. Those who have received breast cancer related surgery, radiotherapy or chemotherapy;
3. Those who are not expected to receive surgery, radiotherapy or chemotherapy related to breast cancer
4. History of other malignant tumors;
5. Pregnant or lactating women;
6. Accompanying active infection and fever;
7. Other serious diseases that may significantly affect clinical trial compliance, such as severe cardiopulmonary dysfunction, liver and kidney dysfunction, poorly controlled diabetes and mental illness.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-08 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
DFS | 1 year；3 years；5 years
  Disease-free survival of patients with locally advanced breast cancer

SECONDARY OUTCOMES:
OS | 1 year；3 years；5 years
  Overall survival of patients with locally advanced breast cancer
Five year survival rate | 1 year；3 years；5 years
  Five year survival rate of patients with locally advanced breast cancer
Local recurrence or distant metastasis rate | 1 year；3 years；5 years
  Local recurrence or distant metastasis rate of patients with locally advanced breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Yan Lin, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Ying Xu, Beijing, China